CLINICAL TRIAL: NCT02475161
Title: A Study to Investigate the Effect of Increased Gastric pH From the Administration of the Proton Pump Inhibitor (PPI) Rabeprazole on the Oral Bioavailability of the Orexin-2 Receptor Antagonist JNJ-42847922 in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Increased Gastric pH on the Oral Bioavailability of the Orexin-2 Receptor Antagonist JNJ-42847922 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107627; 42847922EDI1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Rabeprazole; JNJ-42847922
MeSH Terms: interventions — seltorexant; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNJ-42847922 Plus Rabeprazole (Experimental): Participants will receive JNJ-42847922, 20 milligram (mg) on Day 1 and Day 6. Participants will receive rabeprazole 20 mg once daily from Day 2 to Day 6.
  Interventions: Drug: JNJ-42847922; Drug: Rabeprazole

INTERVENTIONS:
Drug: JNJ-42847922 — JNJ-42847922 will be administered as 20 mg tablet orally.
Drug: Rabeprazole — Rabeprazole will be administered as 20 mg tablet orally.

SUMMARY:
The purpose of this study is to assess the effects of daily administration of rabeprazole on the single-dose pharmacokinetics of JNJ-42847922 in healthy participants.

DETAILED DESCRIPTION:
This is an open-label, single-center, fixed-sequence study designed to assess the effects of multiple oral administration of rabeprazole (a PPI) on the pharmacokinetics of a single oral dose of JNJ-42847922 in healthy participants. The study consists of 3 phases: a Screening Phase of approximately 4 weeks (Days -29 to -2); an Open Label Treatment Phase (Days -1 to 7); and an End-of-Study Phase occurring from 7 to 14 days after the last dose of study drug. All participants will receive JNJ-42847922, orally on Day 1 (alone) and Day 6 (along with rabeprazole).Rabeprazole will be administered orally on Day 2 to Day 6. Pharmacokinetics will primarily be for JNJ-42847922, M12 metabolite and M16 metabolite. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* If a woman, must be postmenopausal (no spontaneous menses for at least 2 years) or surgically sterile (including but not limited to hysterectomy, oophorectomy, salpingectomy, tubal ligation, and tubal occlusion). Women must agree to not donate eggs (ova, oocytes) during the study and for 3 months after the last dose of study drug. Women of child-bearing potential or currently breastfeeding a child are not allowed to participate in the study
* If a man, must agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (BMI) (weight [kilogram {kg}/height^2 [meter]^2) between 18 and 30 kg/m^2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* A participants must be a non-smoker

Exclusion Criteria:

* Current or history of gastrointestinal disorder
* Clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorders, kidney or urinary tract disturbances, significant psychiatric disorder (history of or current diagnosis), history of epilepsy or fits of unexplained black-outs, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, urinalysis, or thyroid stimulating hormone (TSH) at screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication, within 7 days before the first scheduled dose of the study drug (including vitamins and herbal supplements), except acetaminophen and hormonal replacement therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC [0-last]) of JNJ-42847922 | Pre-dose; 10, 20, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours after study drug administration on Day 1 and Day 6
  Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration of JNJ-42847922 will be reported.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-42847922 | Pre-dose; 10, 20, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours after study drug administration on Day 1 and Day 6
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Maximum Observed Plasma Concentration (Cmax) of JNJ-42847922 | Pre-dose; 10, 20, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours after study drug administration on Day 1 and Day 6
  The Cmax is the maximum observed plasma concentration.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC [0-last]) of M12 and M16 | Pre-dose; 10, 20, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours after study drug administration on Day 1 and Day 6
  Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration of M12 and M16.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of M12 and M16 | Pre-dose; 10, 20, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours after study drug administration on Day 1 and Day 6
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Maximum Observed Plasma Concentration (Cmax) of M12 and M16 | Pre-dose; 10, 20, 30, 45 minutes; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours after study drug administration on Day 1 and Day 6
  The Cmax is the maximum observed plasma concentration.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 7 to 14 days after last dose of study drug or early withdrawal)
  An AE was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States